CLINICAL TRIAL: NCT02820974
Title: The Functional Magnetic Resonance Imaging Study on the Processing of Acute Pain and Cognition Among Perimenopause Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC81571656
Record Dates: First submitted 2016-05-12; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Menopause; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy control: Healthy women of child bearing age (25-39) with regular cycles.
- Perimenopause: Women at the age of 40-54 with irregular cycles filling in th criteria of perimenopause.
- Menopause: Women at the age of over 55 without normal cycles filling in th criteria of menopause.

SUMMARY:
There lacks effective early screen system for the migraine-susceptible women during the peri-menopause period. The processing of acute pain and cognition as well as the underling functional magnetic resonance imaging (fMRI) features are suitable for screening pain-susceptible individual. However, there is no study on this issue among the large sample peri-menopause women. The investigators thus designed the current trial to investigate the processing of acute pain and cognition as well as the underling featured functional magnetic resonance imaging (fMRI).The investigators will combine pain behavior,cognitive task, fMRI analysis, psychophysiological interaction (PPI) and suitable statistical package to investigate the relationship between the above mentioned features and the occurrence of migraine and then test the efficacy of these features in predicting migraine development. The investigators will then try to establish the screening system for migraine-susceptible individuals in peri-menopause women.

DETAILED DESCRIPTION:
Although the prevalence of migraine is very high during peri-menopause period, there exist significant individual differences in whether developing migraine among this population. However, there still lacks effective early screen system for the migraine- susceptible women during the peri-menopause period. Individual acute pain processing and its interaction with cognition as well as the underling featured functional magnetic resonance imaging (fMRI) are suitable for screening pain-susceptible individual. Actually, the featured acute pain processing and its interaction with cognition as well as fMRI alterations were reported in two previous small sample trials among pre-menopause population, however, there is no similar study on large sample peri-menopause women. The investigators previously reported abnormal acute pain processing and decreased cognition in the experimental peri-menopause rats as well as peri-menopause women with migraine. The investigators thus raised the current hypothesis that the acute pain processing and its interaction with cognition as well as the underling featured functional magnetic resonance imaging (fMRI) are usable for screening migraine-susceptible individuals among peri-menopause women. In the current project, The investigators will combine pain behavior,cognitive task, fMRI analysis, psychophysiological interaction (PPI) and suitable statistical package to investigated the relationship between the above mentioned features and the occurrence of migraine and then test the efficacy of these features in predicting migraine development. The investigators will then try to establish the screening system for migraine-susceptible individuals in peri-menopause women.

ELIGIBILITY:
Inclusion Criteria:

* 25 years old or above
* Healthy women

Exclusion Criteria:

* Those with history of present illness
* Past history of significant neurological and psychiatric disorders or MRI contraindication

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 years old or above, healthy women from the Department of orthopedics and medical center
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
mean diffusivity | 2-3 days

SECONDARY OUTCOMES:
Acute pain responses represented by Visual Analogue score | 2-3 days
fractional anisotropy | 2-3 days
mean kurtosis | 2-3 days
cerebral blood flow | 2-3 days
functional and structural connectivity | 2-3 days

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hu B, Yu Y, Dai YJ, Feng JH, Yan LF, Sun Q, Zhang J, Yang Y, Hu YC, Nan HY, Zhang XN, Zheng Z, Qin P, Wei XC, Cui GB, Wang W. Multi-modal MRI Reveals the Neurovascular Coupling Dysfunction in Chronic Migraine. Neuroscience. 2019 Nov 1;419:72-82. doi: 10.1016/j.neuroscience.2019.09.022. Epub 2019 Nov 1. PMID 31682827
- [Derived] Hu B, Wang X, He JB, Dai YJ, Zhang J, Yu Y, Sun Q, Lin-FengYan, Hu YC, Nan HY, Yang Y, Kaye AD, Cui GB, Wang W. Structural and functional brain changes in perimenopausal women who are susceptible to migraine: a study protocol of multi-modal MRI trial. BMC Med Imaging. 2018 Sep 6;18(1):26. doi: 10.1186/s12880-018-0272-6. PMID 30189858
- [Derived] Dai YJ, Zhang X, Yang Y, Nan HY, Yu Y, Sun Q, Yan LF, Hu B, Zhang J, Qiu ZY, Gao Y, Cui GB, Chen BL, Wang W. Gender differences in functional connectivities between insular subdivisions and selective pain-related brain structures. J Headache Pain. 2018 Mar 14;19(1):24. doi: 10.1186/s10194-018-0849-z. PMID 29541875